CLINICAL TRIAL: NCT05598177
Title: Effect of Dexmedetomidine Preconditioning on Myocardial Ischemia-reperfusion : a Randomized, Double-blind Clinical Trial
Brief Title: Effect of Dexmedetomidine Preconditioning on Myocardial Ischemia-reperfusion Injury in Patients Undergoing Open Heart Surgery With Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yibin Qin, associate chief physician, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-K125
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Ischemia-Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Experimental): The participant will be infused with dexmedetomidine during anesthesia to protect the myocardium.
  Interventions: Drug: dexmedetomidine
- Group R (Placebo Comparator): The participant will use saline of the same volume as dexmedetomidine as a placebo during anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dexmedetomidine — The participant will pump dexmedetomidine at the rate of 1μg/(Kg·h) for 10 minutes at the beginning of anesthesia induction, and then maintain the pump at a rate of 0.5μg/(Kg·h) during the operation.
  Arms: Group D
Drug: Placebo — The participant will pump saline without dexmedetomidine at the same speed as group D.
  Arms: Group R

SUMMARY:
About 200000 cardiac operations are performed in China every year. Cardiopulmonary bypass is the basic strategy of open-heart surgery, which may lead to myocardial ischemia-reperfusion injury and low cardiac output syndrome. It will inevitably affect the patient's postoperative recovery. A number of studies have shown that dexmedetomidine, as an auxiliary sedative, has the effects of inhibiting stress response, antiarrhythmia and cardiac protection.Dexmedetomidine has been widely used in anesthesia in cardiac surgery. However, at present, few clinical studies pay attention to its mechanism. In this study, dexmedetomidine will be used in cardiac surgery with cardiopulmonary bypass to explore the mechanism of cardiac ischemia-reperfusion injury and the protective effect of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. American Society of Anesthesiologists(ASA) physical status of I-Ⅳ
3. BMI: 18.5-28 kg/m2
4. Type of operation: elective open-heart surgery with cardiopulmonary bypass
5. The patient and/or family members have signed the informed consent.

Exclusion Criteria:

1. Preoperative diagnosis of heart failure 、gradeⅡ-Ⅲ heart block and diabetes
2. LEVF<40%
3. Severe coagulation dysfunction
4. Severe heart, lung, liver and kidney insufficiency
5. Used to have immunosuppressive therapies such as radiotherapy, chemotherapy and glucocorticoid, or have immune system diseases
6. Perioperative allogeneic blood transfusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
troponin T level | before operation
  the level of troponin in the participant's serum
troponin T level | the end of operation
  the level of troponin in the participant's serum
troponin T level | when the participant returned to the ward after the operation
  the level of troponin in the participant's serum
troponin T level | 24 hours after operation
  the level of troponin in the participant's serum
troponin T level | 72 hours after operation
  the level of troponin in the participant's serum

SECONDARY OUTCOMES:
AQP4、iNOS andTNF-α level | before operation
  the level of AQP4、iNOS andTNF-α in the participant's serum
AQP4、iNOS andTNF-α level | when blocking the ascending aorta
  the level of AQP4、iNOS andTNF-α in the participant's serum
AQP4、iNOS andTNF-α level | when developing the ascending aorta
  the level of AQP4、iNOS andTNF-α in the participant's serum
AQP4、iNOS andTNF-α level | when cardiopulmonary bypass is stopped
  the level of AQP4、iNOS andTNF-α in the participant's serum
AQP4、iNOS andTNF-α level | the end of the operation
  the level of AQP4、iNOS andTNF-α in the participant's serum

CONTACTS AND LOCATIONS:
Overall Officials: Yibin Qin, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital Nantong University, Nantong, Jiangsu, China